CLINICAL TRIAL: NCT00828529
Title: A Phase I, Open-label, Randomized Crossover Trial to Investigate the Pharmacokinetic Interaction Between Steady-state Lopinavir/Ritonavir and Single-dose TMC207 in Healthy Subjects.
Brief Title: TMC207-TiDP13-C110: Interaction Study With Lopinavir/Ritonavir in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002545; NCT00980291 (obsolete NCT alias)
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Tuberculosis; HIV
Keywords: TMC207-TiDP13-C110; TMC207-C110; TMC207; Drug-drug interaction; Tuberculosis; HIV; Kaletra; Lopinavir; Ritonavir; Open-label; HIV Infections
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TMC207

SUMMARY:
The purpose of this Phase I, open-label, randomized crossover trial is to investigate the pharmacokinetic interaction between steady-state lopinavir/ritonavir and single-dose TMC207 in healthy volunteers.

DETAILED DESCRIPTION:
TMC207 is being investigated for the treatment of MDR-TB infection. This is a Phase I, open-label, randomized crossover trial in healthy volunteers to investigate the potential interaction between steady-state lopinavir/ritonavir (LPV/rtv) 400/100 mg twice daily and a single dose of 400 mg TMC207. The trial population will consist of 16 healthy volunteers. During 2 sessions, each participant will receive 2 treatments (Treatments A and B) in a randomized order. This means it will be decided by chance if subjects will receive first treatment A, then B or first treatment B, then A.

In Treatment A, participants will receive a single dose of TMC207 400 mg on Day 1. In Treatment B, participants will receive LPV/rtv 400/100 mg twice daily on Days 1 to 24, while on Day 11 a single dose of TMC207 400 mg will be co-administered. The two single doses of TMC207 will be administered 4 weeks apart. Consequently, Treatment B should start 4 days after completion of Treatment A, and Treatment A should start 14 days after completion of Treatment B (counting from the day the last PK sample has been collected). Pharmacokinetic profiles over 336 hours will be determined for TMC207 and its N-monodesmethyl metabolite (M2) after administration of TMC207 400 mg alone (Day 1 of Treatment A), and in combination with steady-state LPV/rtv (Day 11 of Treatment B). Morning predose concentrations of lopinavir and ritonavir will be determined at several time points. Safety and tolerability will be evaluated throughout the trial. Day 1 of Treatment A and on Day 11 of Treatment B, 400 mg TMC207 (1 tablet) will be taken orally in the morning within 10 mins. after completion of a meal. Days 1 to 24 of Treatment B, 2 tablets of Lopinavir/Ritonavir (LPV/rtv = 400 mg lopinavir and 100 mg ritonavir) will be taken in the morning and evening. When LPV/rtv is administered alone, it can be taken with or without food. When co-administered simultaneously with TMC207, LPV/rtv intake will be within 10 mins. after completion of a meal.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Body Mass Index of 18.0 to 32.0 kg/m2, extremes included
* Able to comply with protocol requirements
* Healthy on the basis of a physical examination, medical history, ECG, vital signs and the results of blood biochemistry and hematology test and a urinalysis carried out at screening
* Informed Consent Form signed voluntarily before the first trial-related activity.

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test
* Female, except if postmenopausal since more than 2 years, or posthysterectomy, or post-surgical sterilization
* Hepatitis A, B, or C infection
* Evidence of current use of illicit drugs or opioids or abuse of alcohol
* Currently active or underlying disorders including gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* Any history of significant skin disease or allergy including allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial
* Use of concomitant medication, including over-the-counter products and dietary supplements, except for ibuprofen and paracetamol up to 3 days before the first dose of trial medication
* Recent donation of blood or plasma or participation in a clinical trial
* Subjects with QTc prolongation or any other clinically significant ECG abnormality or a family history of Long QT Syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of steady-state LPV/rtv 400/100 mg twice daily on the pharmacokinetics of TMC207 and its M2 metabolite after single-dose administration of TMC207 400 mg, in healthy volunteers.

SECONDARY OUTCOMES:
The secondary objectives are: to evaluate the effect of single-dose TMC207 on the steady-state plasma concentrations of lopinavir and ritonavir in healthy volunteers; to evaluate the short-term safety and tolerability of co-administration of single-dose

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA

REFERENCES:
- [Derived] Svensson EM, Dooley KE, Karlsson MO. Impact of lopinavir-ritonavir or nevirapine on bedaquiline exposures and potential implications for patients with tuberculosis-HIV coinfection. Antimicrob Agents Chemother. 2014 Nov;58(11):6406-12. doi: 10.1128/AAC.03246-14. Epub 2014 Aug 11. PMID 25114140